CLINICAL TRIAL: NCT03764930
Title: Attention to Retinoblastoma Diagnosed in the Trauma Setting
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, Head of Orbital Diseases and Ocular Oncology, Clinical Professor, Sun Yat-sen University
Other Study IDs: yanghs201812
Record Dates: First submitted 2018-12-01; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Retinoblastoma; Wounds and Injury
MeSH Terms: conditions — Retinoblastoma; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Unsuspected Retinoblastoma — To study the clinical characteristics and treatment outcomes of patients who experienced inadvertent trauma before diagnosis of retinoblastoma.

SUMMARY:
To study the clinical characteristics and treatment outcomes of patients who experienced inadvertent trauma before diagnosis of retinoblastoma.

DETAILED DESCRIPTION:
Retrospective study of the clinical characteristics and treatment outcomes of patients who experienced inadvertent trauma before diagnosis of retinoblastoma and to alert ophthalmologists to the possibility of RB in children presenting with or without trauma-related symptoms and signs.

ELIGIBILITY:
Inclusion Criteria:

* The consecutive patients with RB managed at the ocular oncology service of Zhongshan Ophthalmic Center, Sun Yat-sen University, between January 2013 and August 2018.

Exclusion Criteria:

* The patients who didn't have undergone trauma before diagnosis of RB.

Ages: 1 Month to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Those children who experienced accidental ocular trauma with or without brain involvement before diagnosis of unsuspected RB was studied.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Survival Status | between January 2013 and August 2018
  Outcome at last follow-up

SECONDARY OUTCOMES:
Trauma incidence of RB patients | between January 2013 and August 2018
  We reviewed the computerized diagnostic records of consecutive patients with RB managed at the ocular oncology service of Zhongshan Ophthalmic Center, Sun Yat-sen University, between January 2013 and August 2018. The charts of those patients who had undergone trauma before diagnosis of RB were selected. In addition, we identified the preschool-aged children (age 0-6 years) who underwent surgical treatment for ocular trauma at our hospital during the corresponding period. Then, we calculated the incidence of trauma among RB patients.
RB incidence of pre-school patients with trauma history | between January 2013 and August 2018
  We reviewed the computerized diagnostic records of consecutive patients with RB managed at the ocular oncology service of Zhongshan Ophthalmic Center, Sun Yat-sen University, between January 2013 and August 2018. The charts of those patients who had undergone trauma before diagnosis of RB were selected. In addition, we identified the preschool-aged children (age 0-6 years) who underwent surgical treatment for ocular trauma at our hospital during the corresponding period. Then, we calculated the incidence of RB among pre-school patients with trauma history.

CONTACTS AND LOCATIONS:
Overall Officials: Huasheng Yang, MD,PhD, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided